CLINICAL TRIAL: NCT06716632
Title: A Comparative Analysis of Hypocalcemia Incidence in Patients Undergoing Thyroidectomy: Ligasure vs Conventional Ligation of Vessels by Knot Tying
Acronym: THYROIDECTOMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulab Devi Hospital (Other)
Responsible Party: Principal Investigator, Zain Himayoun, Principal Investigator (Post Graduate Resident), University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAMC/IRB/EA 41/2024
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Hypocalcemia After Total Thyroidectomy; Hypocalcemia
Keywords: thyroidectomy; hyocalcemia
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ligasure (Experimental): Ligasure is a bipolar vascular sealing system utilized to achieve effective control of bleeding and create a bloodless surgical environment. It operates by utilizing an electrical current within the frequency range of 2-4 MHz It induces denaturation of collagen and elastin within the vessels and surrounding tissues. The localized tissue temperatures typically range between 60-100°C, facilitating the fusion of collagen and elastin in the vessel walls. This fusion process creates a durable sealed zone without any carbonization and enables hemostasis in vessels with diameters of up to 7 mm
  Interventions: Device: Using Ligasure for heamostasis
- Knot tying (Experimental): Conventional methods of vessel ligation, which involve the use of ties and suture ligatures, have long been employed in most medical centers
  Interventions: Procedure: Use of conventional knot tying technique for heamostasis

INTERVENTIONS:
Device: Using Ligasure for heamostasis — Ligasure is a bipolar vascular sealing system utilized to achieve effective control of bleeding and create a bloodless surgical environment. It operates by utilizing an electrical current within the frequency range of 2-4 MHz It induces denaturation of collagen and elastin within the vessels and surrounding tissues. The localized tissue temperatures typically range between 60-100°C, facilitating the fusion of collagen and elastin in the vessel walls. This fusion process creates a durable sealed zone without any carbonization and enables hemostasis in vessels with diameters of up to 7 mm.
  Arms: Ligasure
Procedure: Use of conventional knot tying technique for heamostasis — Conventional methods of vessel ligation, which involve the use of ties and suture ligatures, have long been employed in most medical centers. While these techniques effectively control bleeding from vessels, they are time-consuming and carry the risk of harming adjacent structures like the recurrent and superior laryngeal nerves.
  Arms: Knot tying

SUMMARY:
This study aims to address the existing gap in knowledge by conducting a comprehensive comparison of the incidence of hypocalcemia in patients undergoing thyroidectomy using Ligasure versus conventional ligation of vessels by knot tying. Additionally, secondary outcomes such as operative time, intraoperative bleeding, length of hospital stay, and postoperative complications will be assessed to provide a holistic understanding of the two surgical approaches.

DETAILED DESCRIPTION:
Thyroidectomy is surgical removal of all or part of the thyroid gland, which is located in the front of the neck. Depending on how much thyroid tissue is removed, thyroidectomy could be classified into Total thyroidectomy, subtotal thyroidectomy, near total thyroidectomy and lobectomy.

In total thyroidectomy, the entire thyroid gland is removed. In thyroid lobectomy, one lobe of the thyroid gland is removed. In Thyroid lobectomy with isthmectomy, thyroid lobe along with the isthmus is removed. In Subtotal thyroidectomy, a small portion of the thyroid gland is left during the surgery. This portion is near the trachea, parathyroid glands and the recurrent laryngeal nerve. Indications for thyroidectomy are thyroid cancer, MNG, solitary thyroid nodule.

Complications of thyroidectomy include hoarseness or change in voice (33.3%), damage to parathyroid glands causing hypocalcaemia (54.4%), wound infection (3.4%), dysphagia (32.8%). Several risk factors may contribute to the occurrence of post-thyroidectomy complications, including age, gender, enlarged gland size, type of thyroid disease, presence of fibrosis and inflammation, extent of thyroidectomy, and lymph node dissection. Among these complications, hypocalcaemia and recurrent laryngeal nerve injury are the most frequently observed.

The superior and inferior parathyroid glands, located near the thyroid gland, play a vital role in calcium homeostasis by producing parathyroid hormone (PTH), which regulates calcium levels in the bloodstream.

Hypocalcemia, characterized by low serum calcium levels. It is a frequent and significant complication of thyroidectomy due to damage, ischemia, or removal of one or more of the parathyroid glands during surgery. It can be categorized into two main types, transient hypocalcemia and permanent hypocalcemia. The primary difference between these two types lies in the duration. Transient hypocalcemia lasts for 3 months after surgery, while permanent hypocalcemia persists for 3 months or longer after surgery.

To minimize the risk of parathyroid gland damage, various surgical techniques have been developed, including the utilization of energy-based devices such as Ligasure. Ligasure has gained popularity in thyroidectomy procedures due to its potential advantages in terms of precision, hemostasis, and reduced operative time.

Ligasure is a bipolar vascular sealing system utilized to achieve effective control of bleeding and create a bloodless surgical environment. It operates by utilizing an electrical current within the frequency range of 2-4 MHz It induces denaturation of collagen and elastin within the vessels and surrounding tissues. The localized tissue temperatures typically range between 60-100°C, facilitating the fusion of collagen and elastin in the vessel walls. This fusion process creates a durable sealed zone without any carbonization and enables hemostasis in vessels with diameters of up to 7 mm.

Conventional methods of vessel ligation, which involve the use of ties and suture ligatures, have long been employed in most medical centers. While these techniques effectively control bleeding from vessels, they are time-consuming and carry the risk of harming adjacent structures like the recurrent and superior laryngeal nerves. In light of the growing demand for time-saving procedures, particularly in high-volume operating theaters where efficient patient turnover is essential, there is a growing interest in devices or techniques that minimize the reliance on conventional knot-tying or suture ligation for achieving hemostasis. This is particularly important to optimise anesthesia time and improve overall efficiency.

According to a recent study, hypocalcemia occurred in 6.7% of individuals who underwent surgery using the Liga Sure method. In a separate study, 32.4% of patients who had surgery utilising the traditional knot tying technique experienced hypocalcemia.

However, despite the increasing use of Ligasure and other energy devices, there is a paucity of research comparing their efficacy in preventing hypocalcemia after thyroidectomy.

Therefore, this study aims to address the existing gap in knowledge by conducting a comprehensive comparison of the incidence of hypocalcemia in patients undergoing thyroidectomy using Ligasure versus the conventional artery forceps/knot tying technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from both genders.
2. Age between 20 years to 50 years.
3. Patients undergoing Total thyroidectomy for benign thyroid disease.

Exclusion Criteria:

1. Patients having pre-operative hypocalcaemia.
2. Patients having malignant thyroid disease.
3. Patients having recurrent thyroid disease.
4. Patients having lobectomy + isthmectomy.
5. Patients having pro-operative calcium supplements.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Zia-ul-Miraj Ahmad Study Director, MBBS,FRCS, Study Director — Gulab Devi Hospital
Locations (1):
- Gulab Devi Hospital, Lahore, Punjab Province, Pakistan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Time Period/Location:Surgical Department, Gulab Devi Hospital, Lahore, from April 2024 to March 2025.
  Methodology:
  Seventy-six patients who underwent thyroidectomy were randomly allocated using lottery method to the LigaSure (38) and conventional knot-tying (38) groups.
Period: Overall Study
Arm/Group | Ligasure | Knot Tying
Started | 38 | 38
Completed | 38 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligasure | Knot Tying | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Customized [Mean (Full Range); unit: years]
  Age | 37.89 [21 to 50] | 39.29 [23 to 50] | 38.59 [21 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 40
  Male | 21 | 15 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Pakistan | 38 | 38 | 76
Hypocalcemia [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hypocalcemia
Time Frame: 2 Days
Measure: Number; unit: participants
Arm/Group | Ligasure | Knot Tying
Number analyzed (Participants) | 38 | 38
participants | 4 | 3

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Ligasure | Knot Tying
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT06716632/Prot_003.pdf
  • Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT06716632/SAP_004.pdf